CLINICAL TRIAL: NCT04791033
Title: Quality of Life After Hysterectomy for Adenomyosis and Other Benign Gynecological Conditions
Brief Title: Quality of Life After Hysterectomy (AdenoQOL)
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Omtvedt, Principal Investigator, Oslo University Hospital
Other Study IDs: 213906
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Adenomyosis; Quality of Life
Keywords: Hysterectomy; Sexual Health; Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adenomyosis: Patients with adenomyosis
  Interventions: Procedure: Hysterectomy
- Other benign gynecological conditions: Patients with other benign gynecological conditions (i.e: myomas, endometriosis).
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Elective procedure with hysterectomy due to benign gynecological condition

SUMMARY:
Adenomyosis is a disease where ectopic endometrial-like glands affect the muscular wall of the uterus. About 70% of women affected by adenomyosis suffer from dysmenorrhea and menorrhagia. A levonorgestrel-releasing intrauterine device (LNG-IUD) is the first-choice treatment of adenomyosis, but is not always sufficiently effective in all women. Those women often end up removing the uterus (hysterectomy).

Hysterectomy is clinically regarded to be an efficient and final treatment of adenomyosis, but pelvic pain may also prevail after removal of the uterus. This study aimes to investigate the short - and long-term impact of hysterectomy on quality of life (QOL) and sexual function in women with adenomyosis, and further to evaluate if there is any difference compared to women that are removing their uterus due to other benign gynecological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal status defined by having had menstruation within the last 12 months, or age < 50 years if amenorrhea due to hormonal treatment
* Hysterectomy planned due to a benign condition
* Able to communicate in Norwegian or English
* Electronic consent given

Exclusion Criteria:

* Age < 18 years, postmenopausal status or no menstrual bleeding for the last 12 months
* Hysterectomy as part of female-to-male transition
* Pelvic organ prolapse as an indication for hysterectomy
* Gynecological cancer suspected at the time of inclusion
* Not able to communicate in Norwegian or English

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A consecutive sample of women that are scheduled for hysterectomy at the study site, who fulfill eligibility criteria, are invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The impact of hysterectomy on health related quality of life assessed by SF-36 sub scale bodily pain | 1 year
  The Short Form Health Survey (SF-36) measures eight sub scales including bodily pain (BP) which in this study is used as primary outcome. The scales ranges from 0-100, a higher score indicates a better quality of life.

SECONDARY OUTCOMES:
The impact of hysterectomy on health related quality of life assessed by SF-36 sub scales | 5 years
  The Short Form Health Survey (SF-36) measures eight subscales. In this study seven sub scales is used as secondary outcomes: Physical functioning (PF), role physical (RP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE) and mental health (MH). The scales ranges from 0-100, a higher score indicates a better quality of life.
The impact of hysterectomy on health related quality of life assessed by SF-36 eight subscales | 5 years
  The Short Form Health Survey (SF-36) measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The scales ranges from 0-100, a higher score indicates a better quality of life.
The impact of hysterectomy on sexual function assessed by FSFI | 1 year
  The Female Sexual Function Index (FSFI) use a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning. To score the measure the sum of each domain score (sexual desire, arousal, lubrication, orgasm, satisfaction and pain) is multiplied by a domain factor and summed to derive a total FSFI score.
The impact of hysterectomy on sexual function assessed by FSFI | 5 years
  The Female Sexual Function Index (FSFI) use a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning. To score the measure the sum of each domain score (sexual desire, arousal, lubrication, orgasm, satisfaction and pain) is multiplied by a domain factor and summed to derive a total FSFI score.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Omtvedt, MD, Principal Investigator — Oslo University Hospital; Tina Tellum, PhD, Study Director — Oslo University Hospital
Locations (1):
- Marianne Omtvedt, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
We will share the values of the quality of life data.
Supporting Information: Study Protocol
Time Frame: The data is planned to be made available within a year after the publication of all results.
Access Criteria: Access will be granted upon request and evaluation of the intended use of the data. The intended use should primarily gain improved patient care and research into quality of life after hysterectomy and a detailed protocol has to be submitted.